CLINICAL TRIAL: NCT07299058
Title: The Effect of a Guessing Game on Fear, Pain, and Emotional State During Blood Collection in Children Aged 6-12
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, İlknur Bektaş, Academic staff, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DokuzEU-7
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Pain; Blood Sampling Procedure; Fear Anxiety
Keywords: pain; fear; emotional state; children
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled experimental trial. There will be one intervention group and one control group. The intervention and control groups will receive a pretest, followed by the planned interventions during the blood draw. The control group will receive routine care. Both groups will receive posttests after the intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: I Wonder What I Am Play
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: I Wonder What I Am Play — I Wonder What I Am: This is a board game designed to help children over the age of four develop mental, cognitive, and language skills. The game consists of colorful cards with objects (animals, objects, vehicles, etc.) and a tool for placing them on the head. This tool begins with placing the object card to be guessed in the appropriate location, unseen by anyone else, and explaining the object's characteristics, followed by questions.
  Arms: Intervention

SUMMARY:
The aim of this study is to evaluate the effects of a guessing game on fear, pain and emotional state during blood collection in children aged 6-12 years.

DETAILED DESCRIPTION:
Invasive medical procedures, particularly blood draws, are among the most common healthcare procedures in which children experience intense fear, pain, and emotional stress. The literature contains numerous studies on distraction interventions designed to improve children's psychological well-being and reduce the traumatic effects of these procedures. However, the majority of these studies have focused on passive distraction techniques (e.g., watching videos or listening to music), with less emphasis on play-based interventions that involve active child participation (Uman et al., 2013; Koller & Goldman, 2012). A meta-analysis by Birnie et al. (2018) demonstrated that distraction and techniques such as hypnosis are effective in reducing pain and anxiety associated with needle injections in children. Distraction-based approaches, in particular, have been reported to divert children's cognitive capacity from directing the procedure, leading to more positive emotional responses. A review of studies conducted in this area in Turkey reveals that methods such as distraction with music (Özdemir & Karakoç, 2017), blowing bubbles (Karaman & Selimen, 2015), and playing with toys have generally been evaluated. However, studies systematically examining play-based distraction practices that utilize children's cognitive functions such as decision-making, choice, and direction in the field of nursing are rare. A randomized controlled trial conducted by Hacettepe University found that a combination of information provision and an active distraction method (a tablet puzzle game) reduced both pain and fear levels in children (p=0.001-0.005) (Isıyel et al., 2023). Randomized controlled trials in the international literature demonstrate that playing video games, virtual reality, or using interactive technology (e.g., tablet games, VR modules) significantly reduces pain and anxiety during blood collection (Inan & Inal, 2019). | However, these studies often utilize passive or semi-passive distraction applications tailored to age, while predictive game designs that focus entirely on one-on-one interaction with the child are rarely featured in the literature. To this end, this study will evaluate the "Effect of a Guessing Game on Fear, Pain, and Emotional State During Blood Collection in Children Aged 6-12."

ELIGIBILITY:
Inclusion Criteria:

* Being between 6 and 12 years of age
* Not having a previous diagnosis of a serious hematological/psychiatric disease
* The child and parent must be willing to participate in the study
* Being able to speak and understand Turkish

Exclusion Criteria:

* Having received sedation, analgesics, or anxiolytic medication during the procedure
* Having a visual/hearing impairment
* Having previously undergone an invasive procedure on the same day

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain assessment will be measured using a pain scale. The scale is scored from 0 to 10. The higher the score, the greater the pain. | Months 1-2 of the study
Fear assessment will be measured using a fear scale. The scale is scored from 0 to 4. Higher scores indicate higher fear. | Months 1-2 of the study
Emotional outlook assessment will be measured using the Emotional State Scale. The scale is scored from 5 to 25. Higher scores indicate higher negative emotional states. | Months 1-2 of the study

IPD SHARING:
Plan to Share IPD: Undecided
After the study is completed, it is planned to be shared in accordance with the permission given by the ethics committee.